CLINICAL TRIAL: NCT06453499
Title: Silent Lumbar Disc Herniation Syndrome
Status: Recruiting | Type: Observational
Sponsor: Noha Khaled Shoukry (Other)
Responsible Party: Sponsor-Investigator, Noha Khaled Shoukry, lecturer, Cairo University
Organization: Cairo University (Other)
Other Study IDs: PCU
Record Dates: First submitted 2024-06-04; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- physical therapy: core stability exercise
  Interventions: Other: Physical therapy

INTERVENTIONS:
Other: Physical therapy — ultrasound for 5 minutes,Tens and hot packs for 20 minutes, back exercise

SUMMARY:
LDH is a common phenomenon that is often described in association with various pathological processes affecting the neuromuscular and locomotor systems. It is not only associated with pathology but it can also be observed in healthy individuals with no evidence of any dysfunction. Since LDH is observed in such a large percentage of healthy subjects, it is probably more appropriate to perceive it as a physiological phenomenon with silent clinical biomechanical changes

DETAILED DESCRIPTION:
An observational study will be conducted on 180 individuals without any back or lower extremity symptoms. Individuals who agree to participate in the study will be divided into 3 groups based on their MRI findings. Group 1 (silent disc herniation group): has LDH and root compression confirmed by the MRI but has no back or lower extremity symptoms. Group 2 (had a history of disc herniation with an improvement of their symptoms after receiving physical therapy intervention): has LDH and root compression confirmed by the MRI but has no back or lower extremity symptoms. Group 3 (control group): absence of LDH and root compression confirmed by the MRI has no back or lower extremity symptoms. The isokinetic peak torque for knee and ankle muscles and the H reflex will be assessed for all the individual investigating the influence of silent LDH on the isokinetic parameters and the H-reflex of the lower extremity may help in better guiding for lower extremity screening to identify individuals at risk for lower extremity injuries. It is hoped that clinicians will incorporate such information to understand the importance of confirming the improvemnt obtained from the physical therapy intervention with an MRI before discharging the patients to reduce the risk of recurrence……………………………………………………………………………..…………………………………………………………………………………………………………………..

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria patients with LDH and root compression with no back or lower extremity symptoms.

Exclusion Criteria:

* Any previous history that would affect the alignment or the motion to lower extremity joints as fractures or surgery.

Any fixed deformity True leg length discrepancy (>5mm). Any medical condition affecting peripheral nerves as diabetes mellitus. Any neuromuscular dysfunction and vestibular disorder.Sacroiliac pain or dysfunction low back pain.

Radicular or referred or radiating pain Previous lower extremity injury

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A convenience sample of 180 adult males with a mean age of 40-50 years will be recruited to participate in the study. Inclusion criteria for the study groups (Group 1 and 2) LDH and root compression with no back or lower extremity symtoms. Inclusion criteria for the control group (Group 3) absence of LDH and root compression, no back or lower extremity symptoms. Exclusion criteria: Any previous history that would affect the alignment or the motion to lower extremity joints as fractures or surgery. Any fixed deformity True leg length discrepancy (>5mm).Any medical condition affecting peripheral nerves as diabetes mellitus.Any neuromuscular dysfunction and vestibular disorder.Sacroiliac pain or dysfunction low back pain.Radicular or referred or radiating pain Previous lower extremity injury
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
MRI of lumbar disc | three months
  presence or absence of disc herniation will be confirmed by MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided